CLINICAL TRIAL: NCT02575625
Title: Fibroscan® Medical Device, Assessment for Non Invasive Diagnosis of Liver Steatosis
Acronym: TRANSTEATOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: Echosens (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHAO2011-FP/TRANSTEATOSE
Record Dates: First submitted 2015-09-30; First posted 2015-10-14 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Liver Steatosis
Keywords: Liver steatosis; Steatohepatitis; Fibroscan
MeSH Terms: conditions — Fatty Liver | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibroscan exam (Experimental): Step 1: feasibility study of the method on 10 healthy volunteers Step 2: diagnosis study on 50 healthy volunteers (25 between 18-30 years-old and 25 between 40-65 years-old) and on 25 patients whom cares including an hepatic biopsy et whom the histological answer is clean steatosis (NAFLD).
  Experimental procedures consist in:
  * Fibroscan measure, preceded by tracking sonography.
  * liver MRI (for substudy about MRI comparison, in step 2)
  * a blood test for biological assessment of liver functions
  Interventions: Device: Fibroscan; Biological: Blood test for biological assessment of liver function; Device: MRI

INTERVENTIONS:
Device: Fibroscan — Three series oh independent measures Measure done with Fibroscan will be preceded by tracking ultrasonography.
Biological: Blood test for biological assessment of liver function — Blood test for biological assessment of liver function
Device: MRI — Liver MRI

SUMMARY:
Hypothesis of this study is the existence of a relation between parameters measured by FibroScan® FS 502 according to our non invasive method and liver steatosis condition.

This proof of concept validation is made up of two steps:

* Step 1: feasibility study of the method on 10 healthy volunteers
* Step 2: diagnosis study on 50 healthy volunteers (25 between 18-30 years-old and 25 between 40-65 years-old) and on 25 patients whom cares including an liver biopsy et whom the histological answer is clean steatosis (NAFLD).

Experimental procedures consist in:

* Fibroscan measure, preceded by tracking ultrasonography.
* liver MRI (for substudy about MRI comparison, in step 2)
* a blood test for biological assessment of liver functions

DETAILED DESCRIPTION:
Diagnosis of liver lipid overload (named liver steatosis), unrelated to alcohol consumption, still mainly based on histological exam of the liver. An histological continuity exists going from clean liver steatosis (Non Alcoholic Fatty Liver Disease, NAFLD) to steatohepatitis with signs of inflammation and tissue fibrosis (Non Alcoholic Steato-Hepatitis, NASH). It's now well-known that disease can evolve to cirrhosis and its complications.

Hypothesis of this study is the existence of a relation between parameters measured by FibroScan® FS 502 according to our non invasive method and liver steatosis condition.

This proof of concept validation is made up of two steps:

* Step 1: feasibility study of the method on 10 healthy volunteers
* Step 2: diagnosis study on 50 healthy volunteers (25 between 18-30 years-old and 25 between 40-65 years-old) and on 25 patients whom cares including an liver biopsy et whom the histological answer is clean steatosis (NAFLD).

Measures on healthy volunteers enable to do an intra-operator reproductibility analysis, a study of an age effect and a search of potential mechanic aging of the liver.

Experimental procedures consist in:

* Fibroscan measure, preceded by tracking ultrasonography.
* liver MRI (for substudy about MRI comparison, in step 2)
* a blood test for biological assessment of liver functions

The final aim of this study is to propose a device enable medical community to do in vivo hepatic rheology observation, highly correlated to liver lipid overload. After industrialization of this innovation, this diffusion could making easier patients follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects - Steps 1 and 2

  * Age between 18 and 65 years old (2 age groups for step 2 : 18-30 et 40-65 years-old)
  * Written inform consent form signed
  * Affiliated to medical insurance
  * Alcohol consumption d'alcool < 20g/j for women, <30g/j for men
* Patients with liver steatosis - Step 2

  * More than 18 years -old
  * Written inform consent form signed
  * Affiliated to medical insurance
  * Patients with clean steatosis confirmed by histological results of a liver biopsy done the previous month
  * Alcohol consumption d'alcool < 20g/j for women, <30g/j for men

Exclusion Criteria:

* Healthy subjects - Step 1

  * Exposure to chemical poisons (solvents, paints, drugs) in the previous 4 weeks
  * Pregnant women, lactating women, and women in age for procreation and without reliable contraception
  * Presence of ascites
  * Person under guardianship
* Healthy subjects - Step 2

  * Exposure to chemical poisons (solvents, paints, drugs) in the previous 4 weeks
  * Pregnant women, lactating women, and women in age for procreation and without reliable contraception
  * Contraindication to MRI
  * Presence of ascites
  * Person under guardianship
* Healthy subjects - Steps 1 and 2

  * Presence of liver tumor or ascites (diagnosed with MRI or ultrasonography)
  * Abnormal liver function tests (increase of transaminases, gammaGT)
* Patients with liver steatosis - Step 2

  * Exposure to chemical poisons (solvents, paints, drugs) in the previous 4 weeks
  * Pregnant women, lactating women, and women in age for procreation and without reliable contraception
  * Contraindication to MRI
  * Presence of ascites
  * liver tumor
  * Serology anti VHC+ or Ag HBs+
  * Infection by HIV
  * Auto-immun hepatitis
  * Genetic hemochromatosis, Wilson disease, lake of alpha-1-antitrypsin
  * Fibrosis or liver cirrhosis at biopsy
  * Person under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Viscosity in Pa.s | One day
  Digital files recorded by medical device will be mathematically processed for extracting elasticity G' and viscosity G'' curves in accordance with the frequency. These curves use to identify the 5 parameters: mu(M), eta(M), alpha, mu(V), eta(V); which describe visco-elasticity variations with frequency thanks to an Matlab algorithm
Elasticity in kPa | One day
  Digital files recorded by medical device will be mathematically processed for extracting elasticity G' and viscosity G'' curves in accordance with the frequency. These curves use to identify the 5 parameters: mu(M), eta(M), alpha, mu(V), eta(V); which describe visco-elasticity variations with frequency thanks to an Matlab algorithm

SECONDARY OUTCOMES:
Reproductibility quantification in arbitrary unit | through study completion, an average of 2 years
  The 5 estimated parameters (which describe visco-elasticity) will be used to quantify the medical device reproductibility
Age in years | through study completion, an average of 2 years
  The 5 estimated parameters (which describe visco-elasticity) and the age oh the healthy volunteers wil be used to study an age effect
Liver signal intensity changes in decibel | through study completion, an average of 2 years
  Adiposis charge will be assessed by measure of liver signal intensity decrease on T1 sequence in phase opposition compared to in phase signal, after correction by iron quantity

CONTACTS AND LOCATIONS:
Overall Officials: Frederic PATAT, MD, PhD, Principal Investigator — CHRU TOURS
Locations (1):
- University Hospital of Tours, Tours, France

REFERENCES:
- See also: Clinical Investigation Center - Technological Innovations — http://cic-it-tours.fr/
- See also: University Hospital of Tours — http://www.chu-tours.fr/